CLINICAL TRIAL: NCT01741181
Title: Vitamin D Supplementation in Patients With Diabetes Mellitus Type 2 and Low 25(OH)D Concentrations: Does it Help to Improve Endothelial Function-The DIMENSION TRIAL
Brief Title: Vitamin D Supplementation in Patients With Diabetes Mellitus Type 2
Acronym: DIMENSION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); National Healthcare Group, Singapore (Other Government)
Responsible Party: Principal Investigator, Rinkoo Dalan, Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DIMENSION-03
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus Type 2; Vitamin D Deficiency
Keywords: 25(OH)Vitamin D; Diabetes mellitus; Endothelial Function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vitamin D Deficiency; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D supplementation (Active Comparator): Vitamin D3 tablets (cholecalciferol)
  Interventions: Drug: Vitamin D supplementation
- Placebo pill (Placebo Comparator): Placebo pill
  Interventions: Drug: Placebo Pill

INTERVENTIONS:
Drug: Vitamin D supplementation — Vitamin D3 marketed by oneNine57
  Other Names: Vitamin D3-Cholecalciferol 1000units per tablet.
  Arms: Vitamin D supplementation
Drug: Placebo Pill — Placebo pill supplied by oneNine 57 imported to Singapore with approval and import licence from HSA.
  Other Names: Placebo
  Arms: Placebo pill

SUMMARY:
Background and Objectives :

The presence of vitamin D deficiency in patients with type 2 diabetes mellitus (T2DM) is associated with an increased risk of cardiovascular disease (CVD). We aim to see whether supplementation of vitamin D in these patients helps to improve the endothelial function (EF) a surrogate marker of CVD risk.

Hypothesis: Vitamin D supplementation in patients with T2DM and low serum 25(OH) D concentrations (<30ng/ml) will improve EF as measured by the Endo-PAT machine by 0.4 units (30% improvement over baseline) and/or will result in a increase of EPCs (CD133+/KDR+) and CD45dim CD34+/KDR.

The investigators will test this hypothesis by comparing 2 groups of T2DM patients randomized to placebo or vitamin D3 for 16 weeks.

Methods:

This is a 16 weeks trial in which 120 T2DM patients will be screened with the aim to recruit 60 T2DM patients with vitamin D deficiency or insufficiency. Out of these 60 patients , 30 patients will be started on vitamin D supplementation and 30 patients will be given a matched placebo. Endothelial function (EF) will be checked before and after supplementation to see a change in EF.

Significance of Project:

If this study shows a significant improvement of EF, it would justify larger scale studies to show that vitamin D supplementation in patients with T2DM mitigates CVD risk and vitamin D supplementation in patients with T2DM and vitamin D deficiency to improve CVD risk.

DETAILED DESCRIPTION:
Overall Aims: Type 2 Diabetes Mellitus (T2DM) is increasingly more prevalent in Singapore and is a high cardiovascular diseases (CVD) risk factor (1,2). The presence of low serum 25(OH)D concentrations (<30ng/ml) has also been classified as an independent predictor of CVD(3,4) and has been seen to be more prevalent in T2DM (5-7). We aim to see whether replacement with vitamin D in these patients helps to mitigate CVD risk. Since endothelial dysfunction is one of the earliest manifestations of CVD and is a very robust surrogate marker, we aim to measure the endothelial function (EF) before and after vitamin D supplementation to evaluate for beneficial impact on this endpoint.

Specific Aims: Although, there are some small scale studies done with a single high dose replacement of vitamin D2/D3, no studies have been done using regular daily supplementation with vitamin D3 and with measurement of EF using the Endo-PAT machine or measurement of endothelial progenitor cells (EPCs).We are doing this pilot study to see whether replacement with vitamin D results in an improvement of EF as measured using the Endo-PAT and estimation of EPCs and some biomarkers as independent established surrogate markers of CVD risk. The estimation of endothelial progenitor cells has been proposed as a surrogate marker of vascular dysfunction and is known to be reduced in patients with cardiovascular risk factors (8). The no. of circulating endothelial cells (CECs) and endothelial microparticles have been seen to be elevated in patients with cardiovascular risk factors and DM and has also been proposed as a effective surrogate marker. We aim to quantify the no. of endothelial progenitor cells (EPCs) staining positive for CD133+/KDR (kinase insert domain-containing receptor),CD34+/KDR and CD45dim CD34+/KDR , CECs (CD 146+/CD45- ) and EMPs derived from endothelial progenitors (CD45-/CD146+/CD34+/CD117+) and from mature endothelial cells (CD45-/CD146+/CD34+/CD117-).using flow cytometry.

Primary Hypothesis:

Vitamin D supplementation in patients with T2DM and low serum 25(OH) D concentrations (<30ng/ml) will improve EF as measured by the Endo-PAT machine by 0.4 units (30% improvement over baseline) and/or will result in a increase of EPCs (CD133+/KDR+) and CD45dim CD34+/KDR. The investigators will test this hypothesis by comparing 2 groups of T2DM patients randomized to placebo or vitamin D3 for 16 weeks.

Secondary Objectives:

To explore the prevalence of low serum 25(OH) D concentrations (<30ng/ml) in T2DM patients and evaluate the difference in the EF in the two groups. To see whether vitamin D supplementation helps to further improve other parameters such as biomarkers, blood pressure, BMI, urine albumin-to-creatinine ratio (ACR), lipid profile of T2DM patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 Diabetes Mellitus
* HbA1c : 6.0-10.0%
* Male of female aged 21-80 years
* Stable Diabetes, blood pressure and hyperlipidemia medications (a 25% dose adjustment is allowed) in the last three months
* Baseline serum 25(0H)D concentration <30ng/ml for randomisation

Exclusion Criteria:

* Baseline serum 25(OH)D concentration >30ng/ml
* Baseline HbA1c>10.1%
* Baseline hypercalcemia (Ca>2.58 mmol/L)
* Known case of Primary Hyperparathyroidism
* Known to be on bisphosphonates
* Known to be on Vitamin D supplementation of 1000 units daily or more in the last one year.
* Chronic renal failure with eGFR<30ml/min
* Known to have cirrhosis of the liver or transaminitis with ALT/AST >3X ULN
* Patients with h/o sarcoidosis, renal calculi or any malignancy
* Patients on current treatment for tuberculosis
* Pregnancy and Lactation
* Women of childbearing potential not taking effective contraceptive measures.
* Patients on long term glucocorticoids or anti-retroviral drugs
* Patients on orlistat or other over the counter preparations that claim to block fat absorption.
* A change in the type of medications for hypertension, diabetes mellitus and hyperlipidemia in the last three months
* Patients who have undergone any form of bariatric surgery
* Patients known to have any malabsorption disorders
* Patients known to have osteoporosis or of baseline BMD scan shows osteoporosis as T score <-2.5SD (for randomisation)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Endothelial function as assessed by the reactive hyperemia index and endothelial progenitor cells | 16 weeks
  Endothelial function will be tested by using the EndoPAT machine which measures the reactive hyperemia index and by estimating the no. of endothelial progenitor cells in the peripheral blood by flow cytometry.

SECONDARY OUTCOMES:
Markers of endothelial cell activation and thrombogenesis | 16 weeks
  Biomarkers measured include hsCRP, e-selectin,von-willebrand factor(vWF)
No. of circulating endothelial cells and endothelial microparticles | 16-20 weeks
  The no. of circulating endothelial cells and endothelial microparticles will be estimated before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rinkoo Dalan, MBBS, FRCP, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore